CLINICAL TRIAL: NCT03975699
Title: Implications of a Paediatrician-psychologist Tandem for Sickle Cell Disease Care and Impact on Cognitive Functioning
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: 29185057
Record Dates: First submitted 2019-06-04; First posted 2019-06-05 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Sickle Cell Disease
Keywords: paediatric-psychological partnership; child; mental health; integrated care; well-being
MeSH Terms: conditions — Anemia, Sickle Cell; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients in centre 1: Louis-Mourier Hospital: All SCD follow-up consultations were conducted jointly by a paediatrician and a clinical psychologist.
  Interventions: Other: Assessment of psychological repercussions of SCD
- Patients in centre 2: Evry hospital: All SCD follow-up consultations were conducted by a paediatrician alone. The unit had close links with the local psycho-medical paediatric care centre when specialized referrals were necessary.
  Interventions: Other: Assessment of psychological repercussions of SCD
- Patients in centre 3: Clamart hospital: All SCD follow-up consultations were conducted by a paediatrician alone.
  Interventions: Other: Assessment of psychological repercussions of SCD

INTERVENTIONS:
Other: Assessment of psychological repercussions of SCD — Quantitative relevant data culled from medical files and qualitative analysis based on data gathered from child and parent interviews, were collected in the three hospitals.

SUMMARY:
Sickle cell disease (SCD) necessitates a paediatric treatment plan that considers the influence of psychological, family and intercultural factors. At the Louis-Mourier Hospital (APHP) in Colombes, France, a paediatric-psychological partnership where a clinical psychologist accompanies the paediatrician at programmed consultations was introduced.

The psychological repercussions of SCD were assessed among children and their parents treated in Colombes and in two other paediatric units without a paediatric-psychological partnership.

ELIGIBILITY:
Inclusion Criteria:

* Children under 18 years old
* Major form of SCD (SS, SC, Sβ° thal, Sβ+ thal) diagnosed by electrophoresis

Exclusion Criteria:

* Child or parent residing in France less than 6 months
* Having received SCD treatment in more than one centre

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children suffering from SCD and their parents, consulting in one of the 3 hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Rey-Osterrieth complex figure test scores (ROCF recall scores) | 1 day
  The Rey-Osterrieth complex figure test (ROCF) is a neuropsychological assessment in which patients are asked to reproduce a complicated line drawing, first by copying it freehand (recognition), and then drawing from memory (recall). Scoring of drawings is based on the widely used 36-point scoring system (0 being the worst score and 36 the best).

IPD SHARING:
Plan to Share IPD: No